CLINICAL TRIAL: NCT04186507
Title: Indirect Evaluation of Lithium Level in Blood Using Non-invasive Sweat Biosensors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tirat Carmel Mental Health Center (Other Government)
Collaborators: Ariel University (Other)
Responsible Party: Principal Investigator, Anatoly Kreinin, MD, PHD, Head of Psychiatric Department , Clinical Assistant Professor Anatoly Kreinin, MD, PHD, MHA, Tirat Carmel Mental Health Center
Other Study IDs: TiratCarmelMHC
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Lithium Level Detection in Sweat
Keywords: Lithium; Biosensor; Sweat; Major Depressive Disorder; Schizoaffective Disorder; Bipolar Mood Disorder; Schizophrenia
MeSH Terms: conditions — Depressive Disorder, Major; Psychotic Disorders; Bipolar Disorder; Schizophrenia | interventions — Lithium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prelaminary group: To confirm that Li+ is detectable in sweat .
- Spectrophon LTD biosensors for Li+ detection in sweat: In this group will be conducted to estimate the suitability, efficacy and accuracy of developed biosensors for non-invasive detection of Li+ in sweat
  Interventions: Combination Product: Smartwatch with integrated Li+ sensor (provided by Spectrophon LTD)

INTERVENTIONS:
Combination Product: Smartwatch with integrated Li+ sensor (provided by Spectrophon LTD) — To confirm that Li+ is detectable in sweat using Macroduct Sweat Collection System for sweat collection.
  Current studies demonstrate that Li+ can be detected in saliva and in sweat. To confirm it, patients that are on treatment with Li+ will be recruited for this aim; sweat will be collected and checked for Li+ levels.
  To develop the algorithm for Spectrophon LTD biosensors for Li+ levels measurement in sweat that will allow assessing the level of Li+ in blood.
  To evaluate the accuracy and the efficacy of biosensors developed by Spectrophon LTD for Li+ detection in sweat.
  Following positive results in previous objectives, clinical trial will be conducted to estimate the suitability, efficacy and accuracy of developed biosensors for non-invasive detection of Li+ in sweat.
  Other Names: Drug: Lithium
  Groups: Spectrophon LTD biosensors for Li+ detection in sweat

SUMMARY:
Indirect evaluation of the accuracy and the efficacy of biosensors developed for Li+ detection in sweat.

DETAILED DESCRIPTION:
Lithium (Li+) is one of the most widely used and studied medications for treating of Bipolar Mood Disorder, resistant cases of Major Psychiatric Disorders and especially Major Depressive Disorder.

After administration, more than 95% of administered dose of Li+ is eliminated unchanged in the urine, less than 5% - in the saliva, sweat, and feces. Up to 40% of patients that are on Li+ therapy encounter adverse effects that can be explained by drug involvement in various biochemical processes. Li+ efficacy and side effect manifestation are obviously determined by the drug concentration in blood. The optimal way to prevent manifestation of side effects is to control that Li+ serum level is within therapeutic range. A blood test is often ordered to monitor the serum level of Li+ to ensure target serum levels are reached. The available methods for blood Li+ are invasive, time consuming, and cause of discomfort for patients, yet are of a great importance as levels of drug in blood outside the therapeutic range may dramatically affect patient health. It is especially of importance for Li+ treatments it has a narrow therapeutic window - 0.6-1.5 mmol/L. Thus, there is a growing need for a reliable, comfortable, and inexpensive method for detection of Li+ in blood that can be performed easily in an in-patient setting and automatically whenever necessary without the need for a clinic visit out-patient setting.

Spectrophon LTD has developed an algorithm that allows calculation of levels of various compounds contained in sweat using standard PPG sensors with special coating and thus to estimate the levels of corresponding chemicals in the bloodstream. This algorithm has proven useful and accurate in clinical trials on detection of dehydration level, blood sodium level, and blood glucose level. We suggest that Spectrophon biosensors can be used to detect the levels of Li+ in sweat that will allow non-invasive estimation of the level of corresponding medication in blood in real-time.

ELIGIBILITY:
Inclusion Criteria:

* Meeting Diagnostic and Statistical Manual 5th edition (DSM-V) criteria for MDD, BMD, Schizoaffective Disorder, Schizophrenia;
* Patients must be on constant Li+ treatment or prior their first drug administration.
* Ability and willingness to sign an informed consent form for participation in the study.

Exclusion Criteria:

* Evidence of serious disorder;
* Unstable chronic disease;
* Kidney disease
* Pregnancy;
* Contraindication for Li+ treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric Inpatients with MDD, BMD, Schizoaffective Disorder, Schizophrenia.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Lithium sweat concentration | 6 month
  Smartwatch with integrated Li+ sensor (provided by Spectrophon LTD) will be placed on the right wrist of each participant for a non-invasive measurement of blood Li+ level.

CONTACTS AND LOCATIONS:
Locations (1):
- Tirat Carmel Mental Health Center, Tirat Carmel, Haifa District, Israel

IPD SHARING:
Plan to Share IPD: Undecided